CLINICAL TRIAL: NCT05534737
Title: Clinical Trial on the Effectiveness of the Model of Centered Care in the Person in the Geriatric Innovative Actions to Advance in the Change of Model Towards Comprehensive and Person-centered Care. AICP.Com
Brief Title: Clinical Trial on the Effectiveness of the Model of Centered Care in the Person in the Geriatric Population at Home(Project AICP.Com)
Acronym: AICPcom
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not carried out
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 216/2022
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Geriatric Care

STUDY DESIGN:
Intervention Model Description: Randomized, open, multicenter clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Comprehensive and Person-Centered Care Model (AICP Model) +regular assistance from social services
  Interventions: Other: MAICP + usual care of social services
- Control (Other): regular assistance from social services
  Interventions: Other: Control

INTERVENTIONS:
Other: MAICP + usual care of social services — The intervention consists of applying a MAICP from the municipal social services involved for 2 years (summer 2022-summer 2024). To this end, the AICP.com project will sign the necessary institutional agreements to contract and integrate, in the municipal Social Services of each territory, an intervention team that will work with them in a coordinated manner, although its specific task is the implementation of the MAICP during the intervention period of the project and the baseline, intermediate and final evaluations of the effectiveness of this model in the study population.
  Arms: Intervention
Other: Control — usual care of social services
  Arms: Control

SUMMARY:
It is an individualized care model and therefore difficult to define in a concrete way: it is based on respect for the individual characteristics of each person (their beliefs, values, preferences, life history, projects, goals...) to find the available family, social and community resources that best suit them in order to promote their autonomy, their quality of life and their emotional well-being.

The design of the randomized clinical trial proposed here is an external collaboration, not financed, which is adapted to the aforementioned project in its community setting and does not affect it beyond the qualification of the definition of the clinical variables of interest without modifying its original design. With it, it seeks to increase the emerging body of published scientific evidence in favor of carrying out this type of community and primary health care interventions that are centered on the person.

DETAILED DESCRIPTION:
The project consists of a set of complementary actions that are considered convenient for the implementation and validation of the Comprehensive and Person-Centered Care Model (MAICP) and is aimed at elderly people in a situation of dependency or loneliness in two areas of action: homes and homes in their community settings.

The MAICP is articulated on two axes: placing the person at the center while the other elements revolve around them, and organizing support and care in a coordinated manner so that they are offered to the person in their community environment in an integrated manner and that This is not the one that must adapt to the uncoordinated and fragmented existing services. Specifically in the community environment (population at home), the objective is the articulation and coordination of both formal public services, as well as existing community and proximity resources in each environment to encourage older people to continue living at home and in their community in decent conditions, avoiding institutionalization and without burdening families. Work will be done in close collaboration with community social services so that they appropriate the elements and techniques proposed by the model at the end of the project. In it, methodologies such as community intervention, case management, life history and care plans and support for the life project will be articulated, through a professional relationship that promotes good care and maintenance of the dignity of people and their rights, as well as their autonomy to maintain control of their lives. The synergies and use of existing resources in each environment will affect the effectiveness of the MAICP.

ELIGIBILITY:
Inclusion Criteria:

1. Situation of Fragility (defined as social vulnerability by Social Services, based on a global qualitative assessment: loneliness, low level of education or resources, home conditions...) or recognized dependency, who live alone and who do not meet criteria for the third group.
2. Recognized dependency (classified as grade I, II or III according to the Dependency Law based on autonomy for basic activities measured by the Barthel scale and cognitive impairment according to Pfeiffer) who have cohabitants and who do not meet the criteria for the third group.
3. Dependence recognized grade II or III that also meet criteria of clinical complexity, at least 2 major criteria and 1 minor:

Major Criteria: polypharmacy >4 active prescription drugs, >=2 visits to the emergency room last year, >=1 hospital admission in the last year Minor criteria: diagnosis of heart failure, COPD, dementia, and/or Liver disease / diabetes mellitus / osteoarthritis (2 of these 3).

Exclusion Criteria:

* those people who during the baseline period (summer 2022) present an event at the end of follow-up (see Variables) will be excluded.

Relatives or partners of other participants who have already been recruited for meeting inclusion criteria will also be excluded, with the most dependent person being the one with priority for inclusion in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment (<23-65%- score in the MEC test of Lobo -see later Scales of social and health evaluation- evaluated in the first visit) | Up to 2 years
Hospital emergency visits in the last year (up to the date of inclusion, the information will be collected through the contribution of the report or by anamnesis of the participant or caregiver) | Up to 2 years
  Number of visits
Hospital admissions in the last year (up to the date of inclusion, the information will be collected through the contribution of the report or by anamnesis of the participant or caregiver) | Up to 2 years
  Number of admissions
Quality of life/emotional well-being scales, according to cognitive impairment (by MEC result): | Up to 2 years
  Qualid scale (10)The average administration time of the questionnaire is 5 minutes. It has 11 items referring to observable behaviors, indicative of his individual experience with respect to his QoL. They include observation of subjective and affective states of patients
Quality of life/emotional well-being scales, according to cognitive impairment (by MEC result): | Up to 2 years
  CASP-12 scale (Control, Autonomy, Pleasure and Self-realization) is a shortened version of the original CASP-19 scale for quality of life in people aged 65-74 years. is self-administered and consists of 12 items, comprised of 4 areas (Control, Pleasure, Autonomy and Self-actualization), which are evaluated using a 4-point Likert-type scale.
No cognitive impairment (MEC-Lobo >23 - 65%, The WHO-5 scale (12)(WHO-5 in its original version) | Up to 2 years
  evaluates emotional well-being through 3 aspects: positive mood, vitality and general interest. It is a self-administered questionnaire with 5 Likert-type questions (0-5 points), with 0 being the lowest score (less emotional well-being) and 25 the highest (more emotional well-being).
MEC (Mini-Cognitive Examination) by Lobo 1999 (9). The maximum total score is 35 points (cognitive impairment is considered if the score is <23 points) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Castillo, Murcia, Spain